CLINICAL TRIAL: NCT06336642
Title: Structured Personalized Oxygen and Supportive Therapies for Dyspnea in Oncology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0933; NCI-2024-02452 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-03-20; First posted 2024-03-29 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: SPOT-ON (Experimental): Participants will work with the healthcare team to find the best ways to reduce your shortness of breath by finding what combination of treatments work for participant. Participants will receive education about shortness of breath by the research staff in addition to information about standard treatments or medications for your shortness of breath that would be offered by your medical team.
  Interventions: Behavioral: SPOT-ON Early Start; Behavioral: SPOT-ON Delayed Start
- Group 2: SPOT-ON Waitlist (Experimental): Participants will work with the healthcare team to find the best ways to reduce your shortness of breath by finding what combination of treatments work for participant. Participants will receive education about shortness of breath by the research staff in addition to information about standard treatments or medications for your shortness of breath that would be offered by your medical team.
  Interventions: Behavioral: SPOT-ON Early Start; Behavioral: SPOT-ON Delayed Start

INTERVENTIONS:
Behavioral: SPOT-ON Early Start — Participants will start treatment within 3 days of enrollment, which may include: receiving information on breathing techniques, relaxation techniques, posture techniques, and distraction techniques, and/or trying different oxygen-based therapies, such as high-flow nasal cannula, low-flow supplemental oxygen, and non-invasive ventilation with a respiratory therapist.
Behavioral: SPOT-ON Delayed Start — Participants will start treatment within 3 days of enrollment, which may include: receiving information on breathing techniques, relaxation techniques, posture techniques, and distraction techniques, and/or trying different oxygen-based therapies, such as high-flow nasal cannula, low-flow supplemental oxygen, and non-invasive ventilation with a respiratory therapist.

SUMMARY:
To learn about the effect of Structured Personalized Oxygen and Supportive Therapies for Dyspnea in Oncology (SPOT-ON) treatment on the severity of shortness of breath in patients with cancer.

DETAILED DESCRIPTION:
Primary Objectives:

1. To determine the effect of SPOT-ON and Enhanced Usual Care on the change in intensity of dyspnea (NRS) between baseline and 24 h in hypoxemic hospitalized patients with cancer.
2. To determine the effect of SPOT-ON and Enhanced Usual Care on the change in intensity of dyspnea (NRS) between baseline and 24 h in non-hypoxemic hospitalized patients with cancer.

Secondary Objectives:

1. To determine the effect of SPOT-ON and Enhanced Usual Care on patient outcomes over 72 h, including intensity of dyspnea (NRS), unpleasantness of dyspnea (NRS), dyspnea response, ital signs, symptom burden, health-related quality of life (EQ-5D-5L), adverse events, patterns of device use, and hospital outcomes.
2. To identify factors associated with dyspnea response in the SPOT-ON intervention, including patient demographics, preferences, and level of usage of oxygen delivery modalities.
3. To identify patient factors associated with their preferences (after Phase II and Phase III) for each of the oxygen delivery modalities in the SPOT-ON intervention, such as patient demographics and dyspnea characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced cancer (metastatic, locally advanced, recurrent, or incurable).
* Age 18 or older.
* Admitted to a medical floor.
* Dyspnea intensity at rest of at least 4 on a 0-10-point NRS (where 0 = none, 10 = worst).
* Speak English or Spanish.

Exclusion Criteria:

* Hemodynamic instability requiring active Merit Team or ICU team involvement.
* Delirium as per clinical team's assessment in the Electronic Health Record (EHR).
* Severe hypoxemia (SpO2 < 90% despite supplemental oxygen of up to 6 L/min).
* Continuous positive airway pressure (CPAP) use for obstructive sleep apnea, actively using >10 hours a day.
* Respiratory failure necessitating mechanical ventilation (i.e., HFNC or NIV), and planned thoracentesis within 72 hours of enrollment.
* Patients with known pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure: 1.Safety and adverse events (AEs) | [Time Frame: Through study completion; an average of 1 year.]
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hui D, Kim MJ, Thomas S, Sachdev G, Shete S, Rathi N, Hensch N, De La Cruz V, Ontai A, Mahler DA, Li J, Bruera E. Structured Personalized Oxygen and Supportive Therapies for Dyspnea in Oncology (SPOT-ON): A personalized randomized clinical trial protocol. PLoS One. 2025 Dec 2;20(12):e0336691. doi: 10.1371/journal.pone.0336691. eCollection 2025. PMID 41329762
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT06336642/ICF_000.pdf